CLINICAL TRIAL: NCT00003209
Title: A Randomized Phase III Study of Chemotherapy and Radiotherapy Versus Radiotherapy Alone as Adjuvant Treatment to Patients With Node Positive Stages IB or IIA Cervix Cancer
Brief Title: Radiation Therapy With or Without Chemotherapy After Surgery in Treating Patients With Stage IB or Stage IIA Cervical Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Collaborators: Medical Research Council (Other Government)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: EORTC-55954; EORTC-55954; MRC-CE04; COSA; EU-98061; NSGO-CC-9502
Record Dates: First submitted 1999-11-01; First posted 2004-04-14 (Estimated); Last update posted 2012-07-11 (Estimated); Status verified 2012-07

CONDITIONS: Cervical Cancer
Keywords: stage IB cervical cancer; stage IIA cervical cancer; cervical squamous cell carcinoma; cervical adenocarcinoma; cervical adenosquamous cell carcinoma
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Bleomycin; Cisplatin; Fluorouracil; Ifosfamide; Methotrexate; Mitomycin; Vinblastine; Vindesine; Radiotherapy

INTERVENTIONS:
Biological: bleomycin sulfate
Drug: cisplatin
Drug: fluorouracil
Drug: ifosfamide
Drug: methotrexate
Drug: mitomycin C
Drug: vinblastine sulfate
Drug: vindesine
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining chemotherapy with radiation therapy may kill more tumor cells. It is not yet known whether giving radiation therapy with chemotherapy after surgery is more effective than radiation therapy alone after surgery in treating cervical cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of radiation therapy with or without chemotherapy after surgery in treating patients with stage IB or stage IIA cervical cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare relapse free and overall survival after radiation therapy with or without the sequential use of chemotherapy in patients with node positive stage IB or IIA cervical cancer. II. Compare the toxic effects of these two treatments in this patient population. III. Study the effect of the addition of chemotherapy on the pattern of relapse in these patients.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to institution, stage, site of lymph node involvement, parametrial invasion, resection margin status, diameter of the primary lesion, and preoperative brachtherapy. Patients are assigned to one of two treatment arms and begin therapy within 6 weeks of surgery. Arm I: Patients receive radiation therapy to the pelvis with or without brachytherapy and/or para-aortic irradiation for 4-5 weeks. Arm II: Patients receive radiation therapy as in arm I plus 1 of 5 different cisplatin-based combination chemotherapy regimens. The patients preferably receive chemotherapy before radiation therapy, unless doubtful or positive margins are present, then radiation therapy is given first. Regimen I: Cisplatin and fluorouracil are administered on days 1 and 2 of a 21 day cycle. Patients receive 4 cycles of therapy. Regimen II: Bleomycin is administered on day 1 and cisplatin and ifosfamide are administered on day 2 of a 21 day cycle. Patients receive 4 cycles of therapy. The regimen may also be given without bleomycin. Regimen III: Patients receive vindesine on days 1 and 8, cisplatin on day 1, bleomycin on days 2-4, and mitomycin on day 5 (cycles 1 and 3 only). Each cycle lasts 21 days and patients receive 4 cycles of therapy. Regimen IV: Cisplatin and vinblastine are administered on day 1 and bleomycin is administered on days 1, 8, and 15 of a 21 day cycle. Each patient receives 4 cycles of therapy. Regimen V: Patients receive cisplatin and methotrexate on day 1 of each 14 day cycle. Patients receive 6 cycles of therapy. Patients are followed every 3 months for the first 2 years, every 6 months for the next 3 years, then annually for the next 5 years.

PROJECTED ACCRUAL: Approximately 700 patients will be accrued for this study within 4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven stage IB or IIA cervical cancer Squamous cell carcinoma Adenosquamous cell carcinoma Adenocarcinoma Pelvic and/or common iliac or para-aortic lymph node involvement Undergone a radical hysterectomy, complete pelvic lymphadenectomy, and resection of any enlarged common iliac or para-aortic lymph nodes No clear cell carcinoma or small cell carcinoma with neuroendocrine differentiation Resectable disease

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: Not specified Hematopoietic: WBC at least 3500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 14.6 mg/dL Renal: Creatinine no greater than 1.356 mg/dL Creatinine clearance at least 60 mL/min Pulmonary: Maximum breathing capacity at least 30 L/min FEV1 at least 1.0 L No signs of respiratory insufficiency Other: No potentially active site of infection (e.g., fistula or abscesses) No prior or concurrent second malignancy except adequately treated basal cell carcinoma of the skin

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: Not specified Endocrine therapy: Not specified Radiotherapy: No preoperative external radiotherapy Surgery: See Disease Characteristics

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 1997-12; Primary Completion 1999-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jan B. Vermorken, MD, PhD, Study Chair — University Hospital, Antwerp; R. Paul Symonds, MD, FRCP, FRCR, Study Chair — University of Glasgow
Locations (2):
- United Kingdom (2):
  - Derbyshire Royal Infirmary, Derby, England
  - Beatson Oncology Centre, Glasgow, Scotland